CLINICAL TRIAL: NCT04992819
Title: The Effect of Oral Feeding Model With a Chronobiological Approach on Growth Parameters and Discharge Time in Preterm Infants: A Randomized Controlled Study
Brief Title: The Effect of Oral Feeding Model With a Chronobiological Approach in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Ebru Temizsoy, Princiciple İnvestigator, RN, MSc, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25848687
Record Dates: First submitted 2021-07-04; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Breastfeeding; Bottle Feeding; Preterm; Chronobiology Disorders
Keywords: breastfeeding; preterm infants; chronobiological; Human milk; Circadian rhythm; neonate
MeSH Terms: conditions — Breast Feeding; Bottle Feeding; Premature Birth; Chronobiology Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled two groups (control group and experimental group)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Preterm infants in NICU are fed with breast milk and bottle. Although the date is written on expressed breast milk, it is usually not given by checking its suitability for the time of day. Experiment is about labeling breast milk by time of day before giving it to babies. There is no extra intervention during feeding. The breastmilk of the control group patients will be given without matching according to the clinical routine practice.
  Demographic data, anthropometric measurements (weight, height, head circumference of all babies will be recorded in the "Baby Monitoring Form" created by the researcher.
- Chronobiological Approach Nutrition Model (Experimental): Preterm infants in NICU are fed with breast milk and bottle. Although the date is written on expressed breast milk, it is usually not given by checking its suitability for the time of day. The milk of the intervention group patients will be matched circadian and given to the babies. Intervention group's breast milk is labeling by time of day before the each feeding. In the intervention group, a label containing the time of expressed breastmilk will be affixed. Circadian matched milk will be provided at each feeding.
  intervention is;n the intervention group, a label containing the time of expressed breastmilk will be affixed. In the milk preparation room, breast milk will be stored in a separate refrigerator as 08:00-19:59 day milk and 20:00-07:59 night milk.
  Demographic data, anthropometric measurements (weight, height, head circumference of all babies will be recorded in the "Baby Monitoring Form" created by the researcher.
  Interventions: Procedure: Chronobiological Approach Nutrition Model

INTERVENTIONS:
Procedure: Chronobiological Approach Nutrition Model — In the intervention group, a label containing the time of expressed breastmilk will be affixed. In the milk preparation room, breast milk will be stored in a separate refrigerator as 08:00-19:59 day milk and 20:00-07:59 night milk.
  Arms: Chronobiological Approach Nutrition Model

SUMMARY:
As in healthy term babies, the ideal food for preterm infants and sick term babies is breast milk. There are many studies indicating that the composition of breast milk can vary from mother to mother, according to the gestational week of the baby and gender. In new researches on breast milk content; It is argued that breast milk is different during the day and at night, that the micro and macro nutrient content, hormones and some enzymes show different levels of secretion at different times of the day, and that breast milk has a circadian rhythm.

This research is designed as a prospective, randomized, controlled type. The study will be carried out in order to evaluate the effect of Chronobiological Approach Nutrition Model application on baby's growth parameters and discharge time in preterm babies hospitalized in Neonatal Intensive Care Unit (NICU).

Simple randomization method will be used for the study and the babies will be divided into intervention(n=40) and control groups(n=40). The research was carried out with 80 babies followed up in the neonatal intensive care unit.

The milk of the intervention group patients will be matched circadian and given to the babies, the milk of the control group patients will be given without matching according to the clinical routine practice. Demographic data, anthropometric measurements (weight, height, head circumference of all babies will be recorded in the "Baby Monitoring Form" created by the researcher.

DETAILED DESCRIPTION:
Circadian fluctuations in breast milk content are very important in preterm infants fed with expressed breast milk. The composition of breast milk varies throughout the day. In the literature, there is no randomized controlled study suggesting that the breast milk of infants fed with expressed milk should be matched to the baby circadian. In this study, it was aimed to evaluate the effect of Chronobiological Approach Model application on preterm infants growth parameters and discharge time in feeding of preterm infants hospitalized in the neonatal intensive care unit . It is aimed to accelerate the growth of babies by making circadian matching to breast milk in feeding preterm infants and to increase the quality of nursing practices by reducing the length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight >1400 <2500 gram and gestational week ≥32-37 weeks
* Who are feeding only human milk
* Fully enterally fed babies (50-100ml / kg / day)
* Whose parents signed the informed consent to participate in the study were included.

Exclusion Criteria:

* Infants who cannot feed with human milk
* Who receive intravenous fluid, total parenteral nutrition or mixed fluid
* Infants with major congenital, cardiac, respiratory or airway abnormalities and infants who require additional pressure and respiratory support
* Metabolic imbalances, hypoglycemia or electrolyte imbalance
* Narcotic analgesic or sedation therapy
* Whose parents did not sign the informed consent were excluded.

Ages: 32 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2021-07-03 (Actual); Study Completion 2021-07-03 (Actual)

PRIMARY OUTCOMES:
The effect of Chronobiological Approach Nutrition Model application on infants weight gain during circadian matched breastmilk | 30 minute
  Body weight gain- in kilograms
The effect of Chronobiological Approach Nutrition Model application on infants height measured during circadian matched breastmilk | 30 minute
  Height-in meters
The effect of Chronobiological Approach Nutrition Model application on infants head circumference during circadian matched breastmilk | 30 minute
  head circumference-in meters
The effect of Chronobiological Approach Nutrition Model application on infants abdominal circumference during circadian matched breastmilk | 30 minute
  abdominal circumference-in meters

SECONDARY OUTCOMES:
The effect of Chronobiological Approach Nutrition Model application on infant's hospital stay | through study completion, an average of 30 days
  hospital stay- in days
The effect of Chronobiological Approach Nutrition Model application on infant's growth parameters | through study completion, an average of 30 days
  Fenton's growth curves were used for determine percentile level in this research

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Temizsoy, Principal Investigator — Zeynep Kamil Women and Child Diseases Training and Research Hospital. İstanbul, Turkey
Locations (1):
- Zeynep Kamil Women and Child Diseases Training and Research Hospital., Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No